CLINICAL TRIAL: NCT00971776
Title: Voyager I: Patient Discharge Using the AB5000 Portable Driver System
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated due to slow enrollment and change in business priority
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Voyager I: G80013/S001
Record Dates: First submitted 2009-09-02; First posted 2009-09-04 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Acute Cardiac Dysfunction
Keywords: Patient receiving AB5000 ventricle potentially recoverable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: AB Portable Driver System — Evaluate the safety and performance of the AB Portable Driver System in home environment.

SUMMARY:
The AB Portable Driver System will allow patients supported with the Circulatory Support System to be discharged home when their medical condition improves to an ambulating status and will continue to receive the assistance of the AB 5000 ventricle for their heart recovery.

ELIGIBILITY:
Inclusion Criteria:

* The subject is an AB5000 Circulatory Support System patient (in accordance FDA-approved indications for use) who is suffering acute cardiac dysfunction and is potentially recoverable;
* The subject is male or female, age 18 years or older;
* The subject is able to ambulate unassisted;
* The subject is on stable oral anticoagulation over 7 days (INR 2-4) with no active bleeding;
* The subject is willing and able to read, understand and sign the study specific informed consent form;
* The subject agrees to comply with study protocol requirements, including all follow-up visits and completion of Qol and NIH stroke scale assessments.

Exclusion Criteria:

* The subject, pre-device implant, is qualified as a transplant candidate.
* There is an absence of a trained companion.
* There is an absence of a psycho-social support.
* The subject has an inadequate home environment, such as poor access which may hinder movements.
* The subject has experienced hypotension in last 24 hours based on two consecutive readings spaced by 8 hours with systolic blood pressures < 90 mmHg.
* The subject requires respiratory assistance.
* The subject has an active infection (positive blood culture and/or body T ≥ 38 degrees C, and/or WBC ≥ 12K/µL).
* The subject requires tube feeding.
* The subject has any other medical condition requiring hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-06; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Adverse events, Quality of life assessment, NIH Stroke Scale Assessments, and patient outcome after readmission | Pre-discharge, 30 days post-discharge, 90 days or re-admission